CLINICAL TRIAL: NCT07356518
Title: Feasibility and Safety of Incorporating Telehealth Visits Combined With Remote Blood Pressure Monitoring in the Management of Chronic Hypertension in Pregnancy
Brief Title: Telehealth and Remote Blood Pressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00142349
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Hypertension in Pregnancy
Keywords: high blood pressure; pre-eclampsia; hypertension during pregnancy
MeSH Terms: conditions — Hypertension; Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Cycle (Experimental): Participants in this arm will be provided telehealth visits in addition to the blood pressure telemonitoring.
  Interventions: Behavioral: Telehealth visits; Behavioral: In-person visits
- Standard of Care (Active Comparator): In person clinic visits
  Interventions: Behavioral: In-person visits

INTERVENTIONS:
Behavioral: Telehealth visits — remote visits with participants
  Arms: Telehealth Cycle
Behavioral: In-person visits — standard of care visits with care provider in person

SUMMARY:
The purpose of this research study is to compare the management of chronic hypertension during pregnancy using telehealth visits with blood pressure telemonitoring and health coaching as compared to standard in person clinic visits. The study involves pregnant woman aged 18-45 who are receiving care for chronic hypertension. Participation in this research study will last until their baby is delivered. The number of in-person clinic visits depends on the participant's treatment assignment. Those assigned to telehealth visits will have telehealth visits alternating with clinic visits every two weeks until the end of pregnancy week 31. Those assigned to telehealth visits will also have five sessions with a health coach via telephone or video from the time of enrollment until the end of pregnancy week 36.

DETAILED DESCRIPTION:
Hypertension (HTN) in pregnancy requires weekly or bi-weekly in-person visits. Telehealth visits with remote blood pressure (BP) telemonitoring may be an alternative to frequent in-person visits improve adherence. However, the feasibility of this approach in pregnancy is lacking and studies are limited on the use of remote BP telemonitoring in chronic HTN (cHTN) during pregnancy. A digital health platform for BP management in pregnant women at risk for preeclampsia (women with cHTN, prior preeclampsia or kidney disease) found fewer admissions for HTN or suspected preeclampsia in the intervention compared to usual care. There is a critical need to investigate the feasibility (willingness and adherence), and safety of this intervention. Without ascertaining the feasibility of telehealth and remote BP monitoring, it remains a challenge to tackle the no-show rates and suboptimal medication adherence during pregnancy.

Objectives Aim 1: To determine the feasibility of incorporating telehealth clinic visits with remote BP telemonitoring alternating with in-person clinic visits in the management of cHTN in pregnancy in the clinic by evaluating willingness to enroll, completion rate and adherence versus standard care (in-person clinic visits alone). This working hypothesis is that this approach will be as feasible as standard care.

Aim 2: To explore safety outcomes of telehealth clinic visits combined with blood pressure remote telemonitoring alternating with in-person clinic visits in the management of chronic hypertension in pregnant patients in the clinic by measuring the incidence of hypotension, syncope or hospitalization/emergency room visits for severe HTN compared to standard care. The working hypothesis is that this approach will be comparable in safety to standard care.

ELIGIBILITY:
Inclusion Criteria:

* prior diagnosis of Chronic hypertension (cHTN)
* Pregnant women
* Known: documented diagnosis or on antihypertensive medication prior to pregnancy

Exclusion Criteria:

* Any significant chronic medical or psychiatric illness that, in the investigator's opinion, would prevent participation in the study
* Cardiac disorders: cardiomyopathy, angina, Coronary Artery Disease (CAD)
* Current substance abuse disorder
* Multifetal pregnancy
* Participation in another study without prior approval
* Plan to deliver outside Atrium Health Wake Forest Baptist
* Prior stroke
* Severe hypertension
* Suspected or known fetal major structural/chromosomal abnormality or fetal demise

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of telehealth with remote BP telemonitoring compared to standard care | Gestational Week 31
  willingness to enroll (number of patients enrolled divided by number of patients reached), study completion rate, adherence compared to standard care). Adherence will be defined as taking medication at least ≥80% of the time, recording ≥70% of weekly BP readings in the intervention group only and completing ≥70% of antenatal telehealth/clinic visits.
Safety of telehealth combined with telemonitoring compared to standard care | Gestational Week 31
  The number of adverse events reported (hypotension, syncope or hospitalization/emergency room visit for severe HTN

SECONDARY OUTCOMES:
Patient satisfaction Scores | Gestational Week 31
  at the end of 31 weeks, each participant will complete a patient research satisfaction survey - Strongly disagree 0, disagree 1, neither agree nor disagree 2, agree 3, strongly agree 4
Clinical team member (Medical Assistant, Nursing staff, Medical Provider, Scheduler) satisfaction Scores | Gestational Week 31
  at the end of 31 weeks, each provider of record for each participant will be invited to complete a research satisfaction survey. Nurses, medical assistants, schedulers at the Comprehensive Fetal Care Center who have participated in the telehealth visit with remote monitoring will be invited to complete a research satisfaction survey - Strongly disagree 0, disagree 1, neither agree nor disagree 2, agree 3, strongly agree 4

CONTACTS AND LOCATIONS:
Overall Officials: Aderonke O Adeniyi, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article, after de-identification (text, tables and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of data has been approved by an independent review committee identified for this purpose.
  For what types of analysis: to achieve aims of the approval proposal and for individual participant data meta-analysis.
  By what mechanism will data become available: Proposals may be submitted up to 36 months. After 36 months the data will be available in our University's data warehouse.